CLINICAL TRIAL: NCT04146857
Title: Effects of Normobaric Hypoxia on Autonomic Activity During a Nap in Healthy Adults (NAPOXIA)
Brief Title: Autonomic Activity During Nap Under Hypoxia
Acronym: NAPOXIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Anja Maehler, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NAPOXIA
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Hypoxia; Sleep; Healthy
Keywords: Hypoxia; Sleep; Heart rate variability; Sleep architecture
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normoxia (Placebo Comparator): 20.9% oxygen
  Interventions: Other: Normoxia
- Hypoxia 1 (Active Comparator): 15.0% oxygen
  Interventions: Other: Hypoxia 1
- Hypoxia 2 (Active Comparator): 12.8% oxygen
  Interventions: Other: Hypoxia 2

INTERVENTIONS:
Other: Normoxia — Nap in hypoxia chamber at 20.9% oxygen (36 m asl)
  Arms: Normoxia
Other: Hypoxia 1 — Nap in hypoxia chamber at 15.0% oxygen (simulates 2660 m asl)
  Arms: Hypoxia 1
Other: Hypoxia 2 — Nap in hypoxia chamber at 12.8% oxygen (simulates 4000 m asl)
  Arms: Hypoxia 2

SUMMARY:
Sleeping under hypoxic conditions can impair cognition and autonomic nervous activity. A short daytime nap can modify these changes. Here we propose a randomized, cross-over study to evaluate the heart rate variability during a 90 min nap in a normobaric hypoxic chamber. In addition, we will investigate sleep architecture, vigilance, attention and memory.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 25-45 years
* BMI 20 - 28 kg/m^2

Exclusion Criteria:

* Severe, manifest illnesses in need of treatment
* Postoperative phases
* Acute and chronic infections
* Sleep disorders such as sleep apnea, insomnia or somnolence
* Altitude exposure (> 2500 m asl) within 6 months before enrollment
* Regular migraines
* Smoking
* Athletes
* Significant weight change within 1 month before enrollment
* Inability to understand significance and scope of the study
* Drug or alcohol abuse

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | During 90 minutes nap under normoxic (20.9%) vs. 12.8% hypoxic condition
  Mean RR interval measured by polysomnography (ms)

SECONDARY OUTCOMES:
Heart rate variability | During 90 minutes nap under normoxic (20.9%) vs. 15.0% hypoxic condition
  Mean RR interval measured by polysomnography (ms)
Sleep Efficiency (SE) | During 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Measured by continuous polysomnography (min)
Wake After Sleep Onset (WASO) | During 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Measured by continuous polysomnography (min)
Sleep Onset Latency (SOL) | During 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Measured by continuous polysomnography (min)
Low Frequency / High Frequency Band | During 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Mean LF/HF ratio measured by continuous ECG
Standard Deviation 1 / Standard Deviation 2 | During 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Mean SD1/SD2 ratio measured by continuous ECG
RR intervals longer than 50 ms | During 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Percentage pNN50 measured by continuous ECG (%)
Core Body Temperature | During 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Mean temperature measured by continuous double sensor monitoring (°C)
Skin Temperature | During 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Mean temperature measured by continuous double sensor monitoring (°C)
Digit Span Task | After 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Longest memorized digit series (n, normal range 5-9, higher is better)
Psychomotor Vigilance Task Subscale 1 | After 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Number of lapses (normal range 0-6, higher is worse)
Psychomotor Vigilance Task Subscale 2 | After 90 min nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Mean reaction time (normal range 100-500 ms, higher is worse)
Color Stroope Task Subscale 1 | After 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Number of incongruency errors (normal range 0-5, higher is worse)
Color Stroope Task Subscale 2 | After 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Congruent response time (normal range 400-500 ms, higher is worse)
Color Stroope Task Subscale 3 | After 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Incongruent response time (normal range 600-800 ms, higher is worse)
Color Stroope Task Subscale 4 | After 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Congruent accuracy (above 95% is normal, higher is better)
Color Stroope Task Subscale 5 | After 90 minutes nap under normoxic (20.9%) vs. two hypoxic conditions (12.8 and 15%)
  Incongruent accuracy (above 85% is normal, higher is better)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Mähler, PhD, Principal Investigator — Charite University, Berlin, Germany; Alain Riveros, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Experimental & Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of reported articles (text, tables, figures, supplemental data) will be shared after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Result] Riveros-Rivera A, Penzel T, Gunga HC, Opatz O, Paul F, Klug L, Boschmann M, Mahler A. Hypoxia Differentially Affects Healthy Men and Women During a Daytime Nap With a Dose-Response Relationship: a Randomized, Cross-Over Pilot Study. Front Physiol. 2022 May 24;13:899636. doi: 10.3389/fphys.2022.899636. eCollection 2022. PMID 35685284
- See also: Results publication — http://www.frontiersin.org/articles/10.3389/fphys.2022.899636/full